CLINICAL TRIAL: NCT03458637
Title: Lifestyle Intervention of Obese Teenagers (LITE) Program: A Randomized Controlled Trial of Usual Care + LITE Versus Usual Care to Treat Obesity in Children 10-16 Years Who Are Referred to KKH Weight Management Clinic
Brief Title: Lifestyle Intervention of Obese Teenagers (LITE) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Ronald McDonald House Charities Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014441E
Record Dates: First submitted 2017-10-25; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2017-09

CONDITIONS: Adolescent Obesity; Lifestyle Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: One arm will be randomised to usual care The experimental arm group will be randomised to usual care and LITE program
Who Masked: Outcomes Assessor
Masking Description: Staff involved in anthropometric measurements will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LITE Program with usual care. (Experimental): LITE Program with usual care. LITE program involves four x 180 min weekly sessions, followed by three x 90 min monthly sessions, for adolescents and parents. The key aspects covered in the LITE program are in keeping with Health Promotion Board guidelines for the management of overweight and obesity and include healthy food choices and eating patterns, increasing physical activity and reducing sedentary behavior. The parenting aspects aim to support and increase parental capacity to implement and maintain the lifestyle changes.
  Interventions: Behavioral: LITE Program and Usual Care; Behavioral: Usual Care
- Usual Care (Active Comparator): Usual care consisting of Weight management clinic consultation at baseline randomization, 3 and 6 months post randomization in a tertiary setting in KK Hospital. Duration of treatment is 6 months. Qualified pediatrician, trained in screening for causes and medical complications of obesity in children, runs the weight management clinic and review the participant at each visit. Optional physical activity, dietary consultation at each weight management clinic visit.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: LITE Program and Usual Care — Family based lifestyle Intervention
  Arms: LITE Program with usual care.
Behavioral: Usual Care — Usual care consisting of 3 visits to weight management clinic

SUMMARY:
Background: Family-based lifestyle intervention programmes have been known to reduce overweight and improve cardiovascular risk in adolescent obesity [1]. This study was designed to address the gap in service provision of a family based weight management program for overweight and obese adolescents. The LITE (Lifestyle Intervention for obese teenagers) group program is a 6-month, family-based behavioural lifestyle intervention, specifically designed to treat obesity in adolescents 10-16 years referred to the Weight Management Clinic. The main principles underpinning LITE program are that parents are identified as the agents of change responsible for implementing lifestyle change in the family .

Methods: The study design is a two-arm randomized controlled trial that recruited 60 overweight and obese adolescents 10-16 year olds that attended Kandang Kerbau Women and Children's Hospital(KKH) weight management clinic. Adolescents with secondary cause for obesity are excluded. Participants are randomized to LITE program with usual care or usual care.

Briefly, the LITE program involves four x 180 min weekly sessions, followed by three x 90 min monthly sessions, for adolescents and parents. The key aspects covered in the LITE program are in keeping with Health Promotion Board guidelines for the management of overweight and obesity and include healthy food choices and eating patterns, increasing physical activity and reducing sedentary behavior. The parenting aspects aim to support and increase parental capacity to implement and maintain the lifestyle changes. The program takes a solution focused approach with families identifying small changes that they would like to try each week instead of a child-centric approach.

Outcome measurement are assessed at 3 and 6 months post baseline and include anthropometric measurements, physical activity, dietary intake, metabolic profile, improvement in positive parenting behaviour and measurement of family support.

Primary outcome is change in body mass index (BMI) z-score at 6 months. Secondary aim is to evaluate the changes in waist-height ratio and fat percentage change and improvement in positive parenting behaviour.

ELIGIBILITY:
Inclusion Criteria:

* All adolescents aged 10-16 years old who are currently enrolled in the Weight Management Programme

Exclusion Criteria:

* Intellectual disability, significant medical illness that precludes physical activity and significant psychiatric illness
* Secondary cause of obesity
* Taking of medications that can affect weight status
* Poor level of spoken English (adolescent/carer)
* Severe obesity as defined by BMI more than or equal to 40kg/m2
* Sibling who is already participating in the study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 3 months and 6 months
  Investigate the efficacy of LITE + Usual Care in comparison to Usual Care only in reducing BMI-z scores from randomization to 6 months in children 10-16 years of age identified as obese who are referred to the KKH Weight Management Clinic

SECONDARY OUTCOMES:
Body fat percentage | 3 and 6 months
  Investigate the efficacy of LITE + Usual Care in comparison to Usual Care only in reducing body fat percentage from randomization to 6 months in children 10-16 years of age identified as obese who are referred to the KKH Weight Management Clinic
Waist height ratio | 3 and 6 months
  Investigate the efficacy of LITE + Usual Care in comparison to Usual Care only in reducing waist height ratio from randomization to 6 months in children 10-16 years of age identified as obese who are referred to the KKH Weight Management Clinic
Improvement in positive parenting behaviour | 3 and 6 months
  Investigate the efficacy of LITE + Usual Care in comparison to Usual Care only in improvement in positive parenting behaviour from randomization to 6 months in children 10-16 years of age identified as obese who are referred to the KKH Weight Management Clinic. Improvement in positive parenting behaviour is measured using the Parenting Scale which is a 30 item questionnaire administered to a parent to measure dysfunctional discipline styles

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chu Shan Chew, MBBS, Principal Investigator — KK Women's and Children's Hospital

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers based on the informed consent form

REFERENCES:
- [Background] Ho M, Garnett SP, Baur L, Burrows T, Stewart L, Neve M, Collins C. Effectiveness of lifestyle interventions in child obesity: systematic review with meta-analysis. Pediatrics. 2012 Dec;130(6):e1647-71. doi: 10.1542/peds.2012-1176. Epub 2012 Nov 19. PMID 23166346